CLINICAL TRIAL: NCT04900402
Title: Comparison of the Activity Level and Quality of Life of Individuals With Physical Disabilities, Those Who Continue and do Not Continue Rehabilitation During COVID-19
Brief Title: Activity Level and Quality of Life of Individuals With Physical Disabilities
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Fulya Senem Karaahmetoglu, Physiotherapist, Saglik Bilimleri Universitesi
Other Study IDs: continue_rehabilitation
Record Dates: First submitted 2021-05-11; First posted 2021-05-25 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Covid19; Physical Disability; Quality of Life
Keywords: COVİD-19; Activity level; Physical Disabilities; Quality of Life
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with physical disabilities continuing rehabilitation after COVID-19: International Physical Activity Questionnaire Short Form (IPAQ) and Child Quality of Life Scale (PedsQL) questionnaires will be applied to individuals who continue their rehabilitation after the COVID-19 pandemic is declared.
  Interventions: Other: Survey
- Individuals with physical disabilities not continuing rehabilitation after COVID-19: International Physical Activity Questionnaire Short Form (IPAQ) and Child Quality of Life Scale (PedsQL) questionnaires will be applied to individuals who do not continue rehabilitation after the COVID-19 pandemic is declared.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — International Physical Activity Questionnaire Short Form (IPAQ) and Quality of Life Scale for Children (PedsQL)

SUMMARY:
This study; It will be done in order to compare the quality of life and physical activity levels of physically disabled individuals who continue and do not continue rehabilitation during COVID-19. International Physical Activity Questionnaire Short Form (IPAQ) and The Quality of Life Scale for Children (PedsQL) questionnaire will be applied.

DETAILED DESCRIPTION:
Studies on COVID-19, which is spreading rapidly all over the world, show that the pediatric population is less affected than the adult and elderly population. Respiratory complications are the leading cause of death in the chronic neuropediatric population. During the pandemic, rehabilitation staff such as physiotherapists are at risk of transmission and therefore their activities should be suspended. For this reason, a 3-month quarantine was applied for individuals who went to special education and rehabilitation in our country from March 2020 to June 2020, and face-to-face sessions could not be continued in rehabilitation.

The negative effects of social isolation in children and adolescents during the pandemic affect mental and physical health. Studies show the importance of physical rehabilitation for pediatric patients with chronic neurological disorders. Rehabilitation is not continuous; It may cause soft tissue contractures, bone deformities, decline in motor functions, dysphagia and respiratory difficulties, among other complications. Pediatric patients with neurological disorders may also experience decline in motor function. Although it is known that rehabilitation services have started again with the strict implementation of social distance and hygiene rules in our country as of June 2020; while some of the physically disabled individuals continue their rehabilitation, those who do not continue with rehabilitation are at a considerable level. Therefore, our study; it will be made in order to compare the quality of life and physical activity levels of physically disabled individuals who continue and do not continue rehabilitation during COVID-19.

Following the approval of the ethics committee, a questionnaire will be applied to 18 children with physical disabilities who continue rehabilitation and 18 children with physical disabilities but who do not continue rehabilitation during COVID-19. The study will start with the approval of the ethics committee and is planned to be completed in October 2021, within 6 months.

The gross motor levels of the children who meet the inclusion criteria and whose families voluntarily accept to participate in the study are determined according to KMFSS, International Physical Activity Questionnaire Short Form (IPAQ) and Quality of Life Scale for Children (PedsQL) questionnaires will be applied to both children who continue special education and rehabilitation during COVID-19 and children who are not.

ELIGIBILITY:
Inclusion Criteria:

* The consent form informed by their parents was read and signed, Children with physical disabilities between the ages of 2 and 18 (cerebral palsy, spina bifida, down syndrome)
* Level I, II and III, IV and V according to KMFSS,
* The person (child or parent) answering the questionnaire is literate in Turkish,
* Children without mental impairment or with mild and moderate mental impairment will be included, according to the "disabled health committee report" of the hospitals.

Exclusion Criteria:

* Cases who have undergone any surgical operation affecting the trunk and upper extremity and lower extremity in the last six months.
* Children with severe mental impairment will not be included.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with physical disabilities (cerebral palsy, spina bifida, down syndrome etc.)
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of activity level | Baseline
  Measurement of activity level with International Physical Activity Questionnaire Short Form (IPAQ)
Evaluation of quality of life | Baseline
  Measurement of quality of life with Children's Quality of Life Scale (PedsQL)

CONTACTS AND LOCATIONS:
Overall Officials: Fulya Senem KARAAHMETOĞLU, Principal Investigator — Saglik Bilimleri Universitesi; Esra PEHLİVAN, Assoc. Prof., Study Director — Saglik Bilimleri Universitesi; Zeynep Betül ÖZCAN, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Sağlık Bilimleri Üniversitesi, Istanbul, Turkey (Türkiye)